CLINICAL TRIAL: NCT05781581
Title: Main Postoperative Complications After SARS-CoV-2 Infection: A Retrospective Cohort Study
Brief Title: A Retrospective Cohort Study for Main Postoperative Complications After SARS-CoV-2 Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Sichuan Academy of Medical Sciences (Other); Second Hospital of Shanxi Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: retro-MPOC
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Intestines Cancer; Pulmonary Cancer; Liver Cancer; Trauma; Fractures, Bone; Gynecologic Disease
MeSH Terms: conditions — Intestinal Neoplasms; Lung Neoplasms; Liver Neoplasms; Wounds and Injuries; Fractures, Bone; Genital Diseases, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
To explore the relationship between SARS-CoV-2 infection in different time before operation and postoperative main complications (mortality, main pulmonary and cardiovascular complications) 30 days after operation; To determine the best timing of surgery after SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years;
* Patients undergoing any type of surgery in operating room.

Exclusion Criteria:

* Surgery under local anesthesia (without participation of anesthetist)
* Surgery outside the operating room, such as gastrointestinal endoscopy, puncture biopsy, etc
* Patients who cannot determine whether they have had SARS CoV-2 infection before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients having any type of surgery in operating room
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2023-03-19 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 30 days after operation | 30 days after surgery
  All-cause mortality at 30 days after operation

SECONDARY OUTCOMES:
Main pulmonary complications at 30 days after operation | 30 days after surgery
  a composite of postoperative pneumonia, acute respiratory distress syndrome (ARDS) and unexpected ventilation
Major Adverse Cardiovascular Events (MACE) | 30 days after surgery
  a composite of cardiogenic death, myocardial infarction, new-onset heart failure or cardiogenic shock, and cerebrovascular accident (CVA)

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, MD,PHD, Study Chair — Renji Hospital, Shanghai Jiaotong University, School of Medcine